CLINICAL TRIAL: NCT06159894
Title: Implementation of Long-acting Cabotegravir + Rilpivirine Administration Out of "HIV Units".
Acronym: IMAdART
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IMAdART
Record Dates: First submitted 2023-11-14; First posted 2023-12-07 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment with LA CAB + RPV and follow-up at Specialist-Care centers (Specialist-Care arm). (Active Comparator): Treatment with LA CAB + RPV and follow-up at Specialist-Care centers (Specialist-Care arm).
  Interventions: Other: Specialist-Care arm
- Treatment with LA CAB + RPV and follow-up in Polyvalent Day Hospital units (Day Hospital arm). (Experimental): Treatment with LA CAB + RPV and follow-up in Polyvalent Day Hospital units (Day Hospital arm).
  Interventions: Other: DAY HOSPITAL ARM

INTERVENTIONS:
Other: DAY HOSPITAL ARM — The study will evaluate the feasibility and acceptability of the administration of CAB LA + RPV LA as perceived by patients. The focus will be upon both Polyvalent Day Hospital units vs Specialist-Care centers. The evaluations of the two-implementation strategies and their differences will be assessed in essentially descriptive terms.
  The study will also explore the fidelity, uptake and costs of LA CAB + RPV administration upon both Polyvalent Day Hospital units vs Specialist-Care Centers. The utility of the implementation strategies devised to support the delivery LA CAB + RPV out of HIV units/Internal medicine services will also be explored.
  Finally, the study will assess the safety, tolerability and effectiveness LA CAB + RPV administration in Polyvalent Day Hospital units vs Specialist-Care centers in the total sample, as per clinical practice.
  Other Names: acceptability of the administration of CAB LA + RPV LA
  Arms: Treatment with LA CAB + RPV and follow-up in Polyvalent Day Hospital units (Day Hospital arm).
Other: Specialist-Care arm — The study will evaluate the feasibility and acceptability of the administration of CAB LA + RPV LA as perceived by patients. The focus will be upon both Polyvalent Day Hospital units vs Specialist-Care centers. The evaluations of the two-implementation strategies and their differences will be assessed in essentially descriptive terms.
  The study will also explore the fidelity, uptake and costs of LA CAB + RPV administration upon both Polyvalent Day Hospital units vs Specialist-Care Centers. The utility of the implementation strategies devised to support the delivery LA CAB + RPV out of HIV units/Internal medicine services will also be explored.
  Finally, the study will assess the safety, tolerability and effectiveness LA CAB + RPV administration in Polyvalent Day Hospital units vs Specialist-Care centers in the total sample, as per clinical practice.
  Other Names: acceptability of the administration of CAB LA + RPV LA
  Arms: Treatment with LA CAB + RPV and follow-up at Specialist-Care centers (Specialist-Care arm).

SUMMARY:
This is a clinical trial whose main purpose is to evaluate the acceptability of the administration of LA CAB + extended-release RPV as perceived by patients in month 12 in multipurpose day hospital units versus specialized care centers (HIV Units). . Candidates to participate in this study are indicated to receive this medication, so the decision to include the participant in the study will be after the decision to prescribe the drug. These patients will be randomly assigned to one location or another to receive the administration of the medication. Therefore, and after consulting with the AEMPS, it is considered that this is a clinical trial WITHOUT medications. Both the medication and the procedures associated with the follow-up of the participants will follow the usual practice for this type of patient, with the exception of completing the questionnaires aimed at evaluating the primary and secondary objectives of this study.

ELIGIBILITY:
Inclusion Criteria:

* 1. People living with HIV-1 infection; 2. Aged 18 years or older at the time of signing the informed consent. 3. Virologically suppressed (HIV-1 RNA <50 copies/ml) on a stable antiretroviral regimen: i) Documented evidence of plasma HIV-1 RNA measurements <50 copies/mL in the 6 months prior to Screening.

  1. Documented evidence of plasma HIV-1 RNA measurements <50 copies/mL in one determination > 6 months prior to Screening
  2. Documented evidence of plasma HIV-1 RNA measurements <50 copies/mL in one determination < 6 months prior to Screening If the last documented evidence of plasma HIV-1 RNA measurements <50 copies/mL is into the 45 days prior to Screening visit, this determination could replace the screening determination. If all the laboratory results from the Screening Visit are available in the 45 days prior to screening visit, Screening visit and Baseline Visit could be done the same day.

  4. Ability to understand informed consent form and other relevant regulatory documents.

  5. Prior to starting LA CAB + RPV injections, healthcare professionals should have carefully selected patients who agree to the required injection schedule and counsel patients about the importance of adherence to scheduled dosing visits to help maintain viral suppression and reduce the risk of viral rebound and potential development of resistance with missed doses.

  6. Investigators may enrol eligible subjects according to their availability and accessibility.

  7. LA CAB +RPV injection may be preceded by an optional 1-month oral lead-in (OLI) according to the physician's judgement; 8. Participants will be monitored according to usual standard care at their physician's discretion.

  9. Females of child bearing potential will be required to use a highly effective method of contraception. A female, may be eligible to enter and participate in the study if she: i) Is of non-child-bearing potential defined as either post-menopausal (12 months of spontaneous amenorrhea and ≥50 years of age) or physically incapable of becoming pregnant with documented tubal ligation, hysterectomy or bilateral oophorectomy.Female participants who have stopped menstruating for ≥12 months and have <50 years of age but do not have documentation* of ovarian hormonal failure must have a serum FSH test result at screening that is within the post-menopausal range based on the reference provided in the Central Laboratory Manual ii) Note: FSH test in the prior 12 months within the post-menopausal range iii) Is of child-bearing potential with a negative pregnancy test at both Screening and Visit 1 and agrees to use one of the highly effective methods to avoid pregnancy documented

Exclusion Criteria:

* 1. Within 6 months prior to Screening, any plasma HIV-1 RNA measurement ≥50 copies/mL or within the 6 to 12-month window prior to Screening, any plasma HIV-1 RNA measurement >200 copies/mL, or 2 or more plasma HIV-1 RNA measurements ≥50 copies/mL.

  2. Present or past evidence of viral resistance to agents of the NNRTI or INSTI class or prior treatment failure with agents of NNRTI or INSTI class

  3. Any contraindication for LA CAB, LA RPV, oral Cabotegravir or Rilpivirine (see EU SmPC)

  4. Women who are pregnant, breastfeeding or plan to become pregnant or breastfeed during the study

  5. Any evidence of a current Center for Disease Control and Prevention (CDC) Stage 3 disease, except cutaneous Kaposi's sarcoma not requiring systemic therapy, and CD4+ counts <200 cells/µL are not exclusionary.

  6. Participants with moderate to severe hepatic impairment

  7. Any pre-existing physical or mental condition (including substance use disorder) which, in the opinion of the Investigator, may interfere with the participant's ability to comply with the dosing schedule and/or protocol evaluations or which may compromise the safety of the participant

  8. Evidence of Hepatitis B virus (HBV) infection based on the results of testing at Screening for Hepatitis B surface antigen (HBsAg), Hepatitis B core antibody (anti-HBc), Hepatitis B surface antibody (anti-HBs) and HBV DNA as follows: 8.1. Participants positive for HBsAg are excluded; 8.2. Participants negative for anti-HBs but positive for anti-HBc (negative HBsAg status), whether negative or positive for HBV DNA, are excluded 8.3. Note: Participants positive for anti-HBc (negative HBsAg status) and positive for anti-HBs (past and/or current evidence) are immune to HBV and are not excluded.

  9. Asymptomatic individuals with chronic hepatitis C virus (HCV) infection will not be excluded, however Clinicians must carefully assess if therapy specific for HCV infection is required; participants who require or qualify for immediate HCV treatment are excluded(Investigators should consult current treatment guidelines when considering choice of therapy for individuals with chronic hepatitis C virus infection. Participants with hepatitis C virus infection should have undergone appropriate work-up, the chronic hepatitis C infection should not be advanced, and not anticipated to require introduction of new HCV therapy (e.g. with oral direct acting antivirals) during the course of the study).

  10. Unstable liver disease (as defined by any of the following: presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, or persistent jaundice or cirrhosis, or decompensated cirrhosis (eg. ascites, encephalopathy, or variceal bleeding)), known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones or otherwise stable chronic liver disease per investigator assessment)

  11. History of liver cirrhosis with or without hepatitis viral co-infection.

  12. Ongoing or clinically relevant pancreatitis

  13. Ongoing malignancy other than cutaneous Kaposi's sarcoma, basal cell carcinoma, or resected, non-invasive cutaneous squamous cell carcinoma, or cervical and anal intraepithelial neoplasia.

  14. History or presence of allergy or intolerance to the study drugs or their components or drugs of their class. In addition, if heparin is used during pharmacokinetic sampling, participants with a history of sensitivity to heparin or heparin-induced thrombocytopenia must not be enrolled.

  15. Current platelet count<100,000 x109/Land/or those with a current or anticipated need for chronic or systemic anticoagulation or a history of known or suspected bleeding disorder, including a history of prolonged bleeding.

  16. Any evidence of primary resistance based on the presence of any major known Integrase inhibitor (INSTI) or Non-nucleoside reverse transcriptase inhibitor (NNRTI) resistance-associated mutation.

  17. Any verified Grade 4 laboratory abnormality at screening.

  18. Subjects has estimated creatinine clearance <50mL/minute per 1.73 meter square via Chronic Kidney Disease-Epidemiology Collaboration (CKD-EPI) Method

  19. Alanine aminotransferase (ALT) ≥5x ULN, OR ALT ≥3 x ULN and bilirubin ≥1.5 x ULN (with > 35% direct bilirubin).

  20. Treatment with an HIV-1 immunotherapeutic vaccine within 90 days of Screening 21. Use of medications which are associated with Torsade de Pointes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-12-18 (Actual); Primary Completion 2025-04-21 (Actual); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
Acceptability of Intervention Measure (AIM) at M12 | 12 months
  Number and proportion of participants receiving injections with an average composite score greater than or equal to 4 across the questions of Acceptability of Intervention Measure (AIM) at M12

SECONDARY OUTCOMES:
Feasibility of Implementation Measure (FIM) at M12 | 12 months
  Number and proportion of participants receiving injections with an average composite score greater than or equal to 4 across the questions of Feasibility of Implementation Measure (FIM) at M12
FIM and AIM at M3 and M7 | month 3 and month 7
  • Number and proportion of participants receiving injections with an average composite score greater than or equal to 4 across the questions of FIM and AIM at M3 and M7
FIM and AIM at 3, 7 and 12 months | 3, 7 and 12 months
  • Differences among the proportions of participants receiving injections with an average composite score greater than or equal to 4 across the questions of FIM and AIM at 3, 7 and 12 months
FIM and AIM at M3, M7 and M12 answered by patients | 3, 7 and 12 months
  Average composite score across the questions on FIM and AIM at M3, M7 and M12 answered by patients
FIM and AIM answered by HCPs and nonclinical staff at M3, M7 and M12. | 3, 7 and 12 months
  Average composite score on FIM and AIM answered by HCPs and nonclinical staff at M3, M7 and M12.
Number and proportion of patients willing to enroll in the study out of total screened collected at M7 and M12. | Month 7 and Month12.
  Number and proportion of patients willing to enroll in the study out of total screened collected at M7 and M12.
Number and proportion of patients enrolled in the study out of total eligible collected at M7 and M12. | Month 7 and Month12.
  Number and proportion of patients enrolled in the study out of total eligible collected at M7 and M12.
Number and proportion of patients voluntary asking to stop LA CAB+RPV administration out of those enrolled in the Polyvalent Day Hospital units or Specialist-Care centers collected at M7 and M12. | Month 7 and Month12.
  Number and proportion of patients voluntary asking to stop LA CAB+RPV administration out of those enrolled in the Polyvalent Day Hospital units or Specialist-Care centers collected at M7 and M12.
Number and proportion of patients voluntary asking to stop LA CAB+RPV LA administration out of total enrolled in the study collected at M7 and M12. | Month 7 and Month12.
  Number and proportion of patients voluntary asking to stop LA CAB+RPV LA administration out of total enrolled in the study collected at M7 and M12.
Number and proportion of injections occurring within the target window from target date (+/- 7 days of target date) collected at M7 and M12. | Month 7 and Month12.
  Number and proportion of injections occurring within the target window from target date (+/- 7 days of target date) collected at M7 and M12.
WHOQOL-HIV-Bref Questionnaire | Month12
  Average change vs baseline on the seven domains scores derived from WHOQOL-HIV-Bref Questionnaire
HIV Treatment Satisfaction Questionnaire (HIVTSQ) | Month12
  Average change vs baseline on the nine domains scores derived from the HIV Treatment Satisfaction Questionnaire (HIVTSQ)
HIV stigma scale (HSS) | Month 12
  Average change vs baseline on the four domains scores derived from 12-item short version of the HIV stigma scale (HSS)
Average change vs baseline on Preference of CAB+RPV LA injected vs. oral ART | Month 12
  Average change vs baseline on Preference of CAB+RPV LA injected vs. oral ART
Perception of pain and ISRs Questionnaire (PIN) | Month12
  Average change vs baseline on the acceptability domain scores derived from the Perception of pain and ISRs Questionnaire (PIN)
WHOQOL-HIV-Bref questionnaire | Month12
  Changes in domain scores derived from WHOQOL-HIV-Bref questionnaire
HIV Treatment Satisfaction Questionnaire (HIVTSQ) | Month12
  Changes in domain scores derived from HIV Treatment Satisfaction Questionnaire (HIVTSQ)
HIV stigma scale (HSS) | Month12
  Changes in domain scores derived from the short version of the the HIV stigma scale (HSS)
ART preference oral vs LA-injectable and and other aspects related to ART change (FAD questionniare) | Month12
  Changes in utility value derived from ART preference of LA-injected vs oral.
Perception of pain and ISRs Questionnaire (PIN) | Month12
  Changes in the acceptability domain scores derived form value derived from Perception of pain and ISRs Questionnaire (PIN)
Likert scale | Month 7 and Month12.
  Average score of satisfaction on a Likert scale for each implementation strategy used answered by patients, HCPs and nonclinical staff at M7 and M12
Average patient direct resource consumption for the LA CAB + RPV administration in a Polyvalent Day Hospital units and Specialist-Care centers at M3, M7 and M12. | Month 7 and Month12.
  Average patient direct resource consumption for the LA CAB + RPV administration in a Polyvalent Day Hospital units and Specialist-Care centers at M3, M7 and M12.
Number and proportion of people with confirmed HIV-RNA >50 copies/mL | Month12.
  Number and proportion of people with confirmed HIV-RNA >50 copies/mL
Time to LA CAB + RPV discontinuation | Month12
  Time to LA CAB + RPV discontinuation
Frequencies of Adverse Events and Serious AEs | Month12
  Frequencies of Adverse Events and Serious AEs
Design an implementation pathway that can be used as a guide or plan in future sites. | Month12
  If the acceptability of receiving treatment in specialty sites does not differ from receiving it in HIV units or standard hospital settings, the implementation trajectory will include that option in its design or recommendation.

CONTACTS AND LOCATIONS:
Locations (1):
- Fundación Jimenez Díaz, Madrid, Spain